CLINICAL TRIAL: NCT04097015
Title: Using Non-Invasive Electrical Stimulation (NI-ES) to Treat Spinal Cord Injury (SCI)
Brief Title: Using NI-ES to Treat Spinal Cord Injury (SCI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: SCI Research Advancement (Other)
Collaborators: DuBois Vision Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCIRA001
Record Dates: First submitted 2019-09-15; First posted 2019-09-20 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Spinal Cord Injuries; Pain, Neuropathic
Keywords: Electrical Stimulation, Transcutaneous; Spinal Cord Injury; Neutrophic Pain; Functional Movements
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia

STUDY DESIGN:
Intervention Model Description: The intervention model is a single group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): The treatment or intervention is the use of NI-ES using a signal generator, Alpha-Stim M, with an Ocular Interface connected to one channel and a Spinal Interface to the other channel. The treatment is done at home for 40 minutes at a time, twice a day. The upper lids of the closed eyes are treated for 10 minutes and the lower lids of the closed eyes are treated for 10 minutes, alternated throughout the treatment time. The Spinal Interface is placed above the SCI for 40 minutes. The entire procedure is repeated for another 40 minutes for a second time. The participant will treat himself at home.
  Interventions: Device: Alpha-Stim M

INTERVENTIONS:
Device: Alpha-Stim M — Alpha-Stim M with and Ocular Interface and a Spinal Interface

SUMMARY:
NI-ES therapy is a treatment that is being studied to potentially treat pain associated with SCI and may help movement below the injury site.

DETAILED DESCRIPTION:
The overall goal of this study is to assess the use of externally applied micro-current electrical stimulation in a subject with SCI to reduce pain and patient perceived improvement of quality of life first, and second, movement below the SCI injury. The Hypothesis is that NI-ES is beneficial in reducing pain following SCI injury, patient perceived quality of life measures, and functional outcomes. We plan to achieve this goal by conducting a Pain Questionnaire and assessment of movement below the injury site prior to external micro-current electrical stimulation with the Spinal Stim (Alpha-Stim M with the Ocular Interface and the Spinal Interface) and again six weeks following the first treatment. These results will be used to characterize the extent and duration of any improvement in pain and movement as a result of treatment with the Spinal Stim.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* The presence of SCI
* Pain associated with the SCI
* Difficulty with body movement below the SCI

Exclusion Criteria:

* Absence of SCI
* Poor health
* Deemed unsuitable for participation by the Investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-11-18 (Estimated)

PRIMARY OUTCOMES:
Pain reduction measured by Pain Questionnaire | 6 weeks
  Reduce neuropathic pain

SECONDARY OUTCOMES:
Functional movement as measured by the ASIA Motor Score | 6 weeks
  Movement below the SCI

CONTACTS AND LOCATIONS:
Locations (1):
- Home site, Buellton, California, United States